CLINICAL TRIAL: NCT06313723
Title: The Effect of Prenatal Education Given to Pregnant Women Via Podcast During the Non-Stress Test on Maternal Anxiety, Fear and Prenatal Attachment
Brief Title: The Effect of Mother's Anxiety, Fear and Prenatal Connection in the Prenatal Education Given to Pregnant Women Via Podcast During the Non-stress Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YASEMİN AYDIN KARTAL (Other)
Responsible Party: Sponsor-Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBÜ-AYDINKARTAL-030
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Prenatal Education
Keywords: podcast; pregnancy; non-stress testing; fear of birth; prenatal attachment; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind quasi-experimental study
Who Masked: Participant
Masking Description: Single (Participant) Which of the participants is the control or intervention group will be selected by randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (n:52) (Experimental): Pregnant women assigned to the intervention group (52) will be listened to podcasts on a Samsung Galaxy J7 Prime brand phone while undergoing a 20-minute NST procedure.Pregnant women in the intervention group will be made to listen to 3 podcasts consisting of 3 modules lasting an average of 5-6 minutes during the Non-Stress Test. After the podcast is prepared, it will be edited in line with expert opinion and its final version will be given.
  Interventions: Other: Prenatal education management delivered via podcast
- Control group (n:52) (No Intervention): Pregnant women assigned to the control group were given T.R. treatment within the scope of routine care. The Ministry of Health's "Pregnancy and Birth Process" booklet will be given and the pregnant woman's questions will be answered on the topics she wants to get information about.

INTERVENTIONS:
Other: Prenatal education management delivered via podcast — Pregnant women assigned to the intervention group (52) will be listened to podcasts on a Samsung Galaxy J7 Prime brand phone while undergoing a 20-minute NST procedure
  Arms: İntervention group (n:52)

SUMMARY:
This study was planned to determine the effect of prenatal education given via podcast to nulliparous pregnant women who applied to the Non-Stress Test Polyclinic of the University of Health Sciences, Istanbul Bagcilar Training and Research Hospital, on maternal anxiety, fear and fetal attachment. The research, planned in a randomized controlled quasi-experimental design, will be carried out with nulliparous pregnant women (n:104) who apply to the Non-Stress Test polyclinic of the University of Health Sciences Istanbul Bağcılar Training and Research Hospital. Pregnant women who voluntarily participate in the research will be divided into intervention (n: 52) and control (n: 52) groups according to the computer-assisted simple random sampling technique. The intervention group, nulliparous pregnant women, will listen to 3 podcasts of 5-6 minutes. Pregnant women in the control group will be given a booklet on the pregnancy and birth process from the Ministry of Health as part of routine care. "Personal Information Form", "State-Trait Anxiety Inventory", "Wijma Birth Expectation/Experience Scale Version A" and "Prenatal Attachment Inventory" will be applied to all pregnant women included in the study.

DETAILED DESCRIPTION:
This study was planned to determine the effect of prenatal education given via podcast to nulliparous pregnant women who applied to the Non-Stress Test Polyclinic of the University of Health Sciences, Istanbul Bagcilar Training and Research Hospital, on maternal anxiety, fear and fetal attachment. The population of the research will consist of nulliparous pregnant women who applied to the Non-Stress Test polyclinic of the University of Health Sciences Istanbul Bağcılar Training and Research Hospital in 2024. The sample of the research will consist of 104 pregnant women who meet the sample selection criteria and participate in the study. Pregnant women who volunteer to participate in the research will be included in the study. The study will be carried out in two groups: the "intervention group", which receives prenatal education with podcasts, and the "control group", which receives routine care. Computer-assisted randomization will be used in the study, and the number of cases will be entered through the program with the URL address https://www. Random assignment was made to 52) and control (n:52) groups. Consent will be obtained from pregnant women using the "Informed Voluntary Consent Form" before the application. Pregnant women assigned to the intervention group will be given a 20-minute NST procedure while listening to a podcast on a Samsung Galaxy J7 Prime phone. Podcast duration is planned to be 5-6 minutes and 3 podcasts will be listened to. Pregnant women in the control group receive T.R. treatment within the scope of routine care. The Ministry of Health's booklet on pregnancy and birth process will be provided. "Personal Information Form", "State-Trait Anxiety Inventory", "Wijma Birth Expectation/Experience Scale Version A" and "Prenatal Attachment Inventory" will be applied to all pregnant women included in the study. Before the data collection forms are implemented, an "Informed Voluntary Consent Form" will be applied to the participants. State-Trait Anxiety Inventory", "Wijma Birth Expectation/Experience Scale Version A" and "Prenatal Attachment Inventory" will be applied to all groups before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being primigravida
* Speaking and understanding Turkish
* To be literate
* Being a pregnant woman admitted to Istanbul Bağcılar Training and Research Hospital Non-Stress Test outpatient clinic or obstetrics and gynaecology open observation department,
* 24 to 32 weeks of gestation in nulliparous pregnant women
* Singleton pregnancy

Exclusion Criteria:

* Pregnant women diagnosed with high-risk pregnancy
* Fetal-obstetric complement complement (preterm labor, hypertension, diabetes, etc.)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 10 minutes
  Reported based on the literature, the form includes questions regarding socio-demographic data and obstetric characteristics of nulliparous pregnant women. Regarding demographic characteristics, the form includes age, gestational age, education level, income may change, spousal support, spouse and individual baby wish status, prenatal follow-up numbers, pregnancy planning status, prenatal education and information availability and where it was obtained. has been given.
State-Trait Anxiety Inventory(D-SKE) | 10 minutes
  It contains two separate scales: State Anxiety Inventory (SCI) and Trait Anxiety Inventory (SCI), which consist of a total of 40 items. There are two types of expressions in D-SKE. Direct expressions express negative emotions, while reverse expressions express positive emotions. In the DCI, the reverse statements are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. In SCI, reverse statements constitute items 21, 26, 27, 30, 33, 36 and 39. After the total weights of direct and reverse expressions are found separately, the total weight score of reverse expressions is subtracted from the total weight score obtained for direct expressions. A predetermined and unchanging value is added to this number. This unchanged value is 50 for DKE and 35 for SKE. The final value obtained is the individual's anxiety score. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Wijma Birth Expectation/Experience Scale Version A (W-DEQ A) | 10 minutes
  The scale consists of 33 items. The answers on the scale are numbered from 0 to 5 and are in a six-point Likert type. 0 means "completely" and 5 means "not at all". The minimum score that can be obtained from the scale is 0 and the maximum score is 165. It is calculated by reversing items 2, 3, 6, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27, 31 of the scale. It is stated that as the score obtained from the scale increases, the fear of birth experienced by women increases. W-DEQ A scores on the scale; women who have low degree of fear of childbirth (W-DEQ A score ≤37), women who have moderate fear of childbirth (those with W-DEQ A score=38-65), women who have severe fear of childbirth (W-DEQ A score=66-84). ) and those with clinical degree of fear of childbirth (W-DEQ A score ≥85).
Prenatal Attachment Inventory (PBI) | 10 minutes
  PBI was developed to explain the thoughts, feelings and situations experienced by women during pregnancy and to determine the level of attachment to the baby in the prenatal period and consists of a total of 21 items. Each item in the PBI is a four-point Likert-type scale with a score between 1 and 4. In PBI, "Never" is scored as 1, "Sometimes" as 2, "Frequently" as 3, and "Always" as 4. A minimum of 21 and a maximum of 84 points can be obtained from PBI. The increase in the score obtained from the PBI indicates that the attachment level of the pregnant woman also increases.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory(D-SKE) | 10 minutes
  It contains two separate scales: State Anxiety Inventory (SCI) and Trait Anxiety Inventory (SCI), which consist of a total of 40 items. There are two types of expressions in D-SKE. Direct expressions express negative emotions, while reverse expressions express positive emotions. In the DCI, the reverse statements are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. In SCI, reverse statements constitute items 21, 26, 27, 30, 33, 36 and 39. After the total weights of direct and reverse expressions are found separately, the total weight score of reverse expressions is subtracted from the total weight score obtained for direct expressions. A predetermined and unchanging value is added to this number. This unchanged value is 50 for DKE and 35 for SKE. The final value obtained is the individual's anxiety score. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Wijma Birth Expectation/Experience Scale Version A (W-DEQ A) | 10 minutes
  The scale consists of 33 items. The answers on the scale are numbered from 0 to 5 and are in a six-point Likert type. 0 means "completely" and 5 means "not at all". The minimum score that can be obtained from the scale is 0 and the maximum score is 165. It is calculated by reversing items 2, 3, 6, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27, 31 of the scale. It is stated that as the score obtained from the scale increases, the fear of birth experienced by women increases. W-DEQ A scores on the scale; women who have low degree of fear of childbirth (W-DEQ A score ≤37), women who have moderate fear of childbirth (those with W-DEQ A score=38-65), women who have severe fear of childbirth (W-DEQ A score=66-84). ) and those with clinical degree of fear of childbirth (W-DEQ A score ≥85).
Prenatal Attachment Inventory (PBI) | 10 minutes
  PBI was developed to explain the thoughts, feelings and situations experienced by women during pregnancy and to determine the level of attachment to the baby in the prenatal period and consists of a total of 21 items. Each item in the PBI is a four-point Likert-type scale with a score between 1 and 4. In PBI, "Never" is scored as 1, "Sometimes" as 2, "Frequently" as 3, and "Always" as 4. A minimum of 21 and a maximum of 84 points can be obtained from PBI. The increase in the score obtained from the PBI indicates that the attachment level of the pregnant woman also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No